CLINICAL TRIAL: NCT05655728
Title: Efficacy and Safety of Metformin in Alport Syndrome: A Randomized, Double-blind, Placebo-controlled Study in China
Brief Title: Treatment With Metformin in Chinese Children With Alport Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jie DING, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCCAS
Record Dates: First submitted 2022-12-08; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Alport Syndrome; Metformin
MeSH Terms: conditions — Nephritis, Hereditary | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin intervention treatment group (Active Comparator)
  Interventions: Drug: Metformin
- The placebo treatment group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — The participants will receive treatment of metformin (initial dose of 500 mg/day, within 2 weeks reaching the maximum tolerated dose [maximum: 1500 mg/day]).
  Arms: Metformin intervention treatment group
Other: Placebo — The participants will receive treatment of placebo.
  Arms: The placebo treatment group

SUMMARY:
This single-center, prospective, double-blind randomized placebo-controlled trial will evaluate the efficacy and safety of metformin in Chinese children with Alport syndrome who have received (and continue to receive)) ACEi/ARB.

ELIGIBILITY:
Inclusion Criteria:

* (1) The diagnostic of Alport syndrome-hematuria with or without proteinuria meets one or more of the following 4 items: i) Immunofluorescence staining of the α5 (IV) chain of the glomerular basement membrane was abnormal; ii) electron microscopy of renal biopsy showed diffuse changes in the glomerular basement membrane; iii) There was one pathogenic variant in the COL4A5 gene or two pathogenic variants in the COL4A3/COL4A4 gene; iv) Family history of Alport syndrome.

  (2) Age is older than or equal to 10 years old. (3) The 24-hour urine protein quantification was greater than 150mg and the urine microalbumin-creatinine ratio was greater than 30 mg/g.

  (4) The estimated glomerular filtration rate (24-hour creatinine clearance) was greater than 45 mL/min/1.73m2.

  (5) Accept the maximum tolerated dose of renin-angiotensin-aldosterone system blockers (Blood pressure in the clinic was in the 50th percentile of the same age, same sex and same height but greater than 90/60mmHg, blood potassium was normal, and the increase of blood creatinine did not exceed 30%) for at least 3 months.

Exclusion Criteria:

* (1) Vitamin B12 deficiency was uncorrected. (2) Treated with Furosemide, amiloride, and nifedipine. (3) Hypertension, chronic liver disease, chronic heart disease, and chronic kidney disease resulting from causes except Alport syndrome.

  (4) History of hyperlactatemia. (5) Allergy to metformin. (6) kidney transplant. (7) Poor compliance. (8) Type 1 diabetes.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-01-03 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy of metformin for Alport syndrome | 24 months
  either decrease in proteinuria or steady eGFR from baseline. To assess the decrease in proteinuria or steady eGFR from baseline to month 12 or month 24 under metformin treatment compared to placebo
Safety of metformin for Alport syndrome | 24 months
  The occurrence of adverse events. Safety will be assessed by monitoring adverse drug events, physical examinations and clinical laboratory test through 24 months

IPD SHARING:
Plan to Share IPD: No